CLINICAL TRIAL: NCT01146522
Title: A Multiple-dose, Parallel Group Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LCQ908 in Patients With Severe Hypertriglyceridemia and Chylomicronemia (Phenotypes I and V)
Brief Title: Safety, Tolerability,Pharmacokinetics(PK)and Pharmacodynamics(PD)Assessment of LCQ908 in Patients With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCQ908A2212
Record Dates: First submitted 2010-06-09; First posted 2010-06-17 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-12

CONDITIONS: Hyperlipoproteinemia
Keywords: Familial hyperchylomicronemia; Lipoprotein lipase deficiency; Hyperlipoproteinemia; Triglycerides; Hypertriglyceridemia; LCQ908; Hyperlipoproteinemia associated with lipoprotein lipase deficiency
MeSH Terms: conditions — Hyperlipoproteinemias; Hyperlipoproteinemia Type I; Hypertriglyceridemia | interventions — pradigastat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LCQ908 (Experimental)
  Interventions: Drug: LCQ908
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCQ908
  Arms: LCQ908
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess safety, tolerability, and effect of LCQ908 on blood lipids in patients with severe hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hyperlipoproteinemia Type I or Type V willing and medically able to discontinue their lipid lowering medication (if prescribed).
* Non breast feeding women.
* Women of child bearing potential practicing appropriate contraception with a negative pregnancy test before dosing.

Exclusion Criteria:

Patients with:

* uncontrolled type 1 or type 2 diabetes mellitus,
* active pancreatitis (the month prior to study start),
* history of drug or alcohol abuse within the 12 months prior to dosing,
* or any surgical or medical condition, acute or unstable chronic disease which may, based on the investigator's opinion, jeopardize the patient in case of participation in the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial plasma triglycerides | baseline and 3 weeks after initiation of each dose level (a test meal will be served at baseline and on Day 21 of treatment)

SECONDARY OUTCOMES:
Blood concentration to characterize LCQ908 kinetics | serial blood samples will be collected from all patients enrolled in the study on Day 21 of treatment with each dose
Different blood lipid biomarkers (such as phospholipids, apolipoproteins, and free fatty acids) | after 3 weeks of treatment with each dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Québec, Canada

REFERENCES:
- [Derived] Meyers CD, Tremblay K, Amer A, Chen J, Jiang L, Gaudet D. Effect of the DGAT1 inhibitor pradigastat on triglyceride and apoB48 levels in patients with familial chylomicronemia syndrome. Lipids Health Dis. 2015 Feb 18;14:8. doi: 10.1186/s12944-015-0006-5. PMID 25889044
- See also: Results for CLCQ908A2212 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7263